CLINICAL TRIAL: NCT00535860
Title: A Multicenter, Randomized, Parallel Study to Assess the Clinical Efficacy, Safety, and Tolerability of ViaDerm-hPTH (1-34) in Comparison to Subcutaneous Injection of Forteo in Postmenopausal Women With Osteoporosis
Brief Title: Efficacy & Safety of ViaDerm-hPTH(1-34) Compared to Forteo SC in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TransPharma Medical (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Efrat Kochba, TransPharma Medical Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS 82-000-04; I2Y-MC-GHFE
Record Dates: First submitted 2007-09-25; First posted 2007-09-26 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Transdermal; hPTH(1-34)
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 50 mcg (Experimental): ViaDerm transdermal delivery
  Interventions: Drug: Teriparatide
- 80 mcg (Experimental): Add Via-Derm transdermal delivery
  Interventions: Drug: Teriparatide
- 20 mcg (Active Comparator): Subcutaneous injection
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide — Daily for 96 days
  Other Names: Forteo; Forsteo; LY333334

SUMMARY:
The purpose of this study is to assess the clinical efficacy, safety, and tolerability of ViaDerm-shPTH [1-34] transdermal delivery in comparison to subcutaneous injection of rhPTH[1-34] following 3-month treatment in postmenopausal women with Osteoporosis

ELIGIBILITY:
Main Inclusive Criteria:

* Post-menopausal women aged between 55 to 85 years (inclusive)
* Posterior-Anterior lumbar vertebral and/or femoral neck BMD T-score by DXA ≤-2.5 SD.
* Have normal serum PTH, thyroid stimulating hormone (TSH) (only for patients treated with thyroid hormone), and prolactin values.

Main Exclusive Criteria:

* Subjects who have a clinical significant or unstable medical or surgical condition that may preclude safe and complete study participation
* Current diagnoses of disorders known to affect bone metabolism including hyperthyroidism, hyperparathyroidism, osteomalacia, or Paget's disease
* Prior osteoporosis treatment with fluoride or strontium at any time; or any IV treatment with bisphosphonates in the past or oral bisphosphonate for more than 1 month in the past 24 months prior to randomization.
* Any condition or disease that may interfere with the ability to have, or to evaluate a DXA scan

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint 96 days in procollagen 1 N-terminal propeptide (P1NP) | Baseline, 96 days

SECONDARY OUTCOMES:
Change from baseline in C-terminal telopeptide of type I collagen (CTX-1.) | Baseline, 96 days
hPTH (1-34) Pharmacokinetic AUC of ViaDerm-hPTH (1-34) and teriparatide SC. | Baseline, 96 days
Ratio of hPTH (1-34) AUC of transdermal treatment and subcutaneous injection | Baseline, 96 days
Ratio of hPTH (1-34) Cmax of transdermal treatment and subcutaneous injection | Baseline, 96 days
hPTH (1-34) Pharmacokinetic Cmax of ViaDerm-hPTH (1-34) and teriparatide SC. | Baseline, 96 Days
Percentage of patients with serum total calcium above the upper limit of normal range | Over 96 days
Percentage of patients with serum total calcium more than 1 mg/dl above the upper limit of normal range | Over 96 days
Number of participants with hPTH (1-34) specific antibody immune response | Baseline, 96 days
Draize score for erythema and edema | Over 96 Days
Visual Analog Scale (VAS) pain assessment | Over 96 days

CONTACTS AND LOCATIONS:
Overall Officials: Efrat Kochba, MD, Study Director — TransPharma-Medical Ltd.
Locations (10):
- Czechia (2):
  - Osteocentrum FN, Hradec Králové
  - Osteocentrum 3 .Interni Klinika 1. LFUK a VFN, Prague
- Hungary (5):
  - Drug Research Center, Balatonfüred
  - Semmelweis University Department of Orthopedic, Budapest
  - Kenezy Gyula Hospital Department of Rheumatology, Debrecen
  - Szent Andras Hospital-Heviz, Hévíz
  - Szent Ferenc Hospital Department of Rheumatology, Miskolc
- Israel (3):
  - Hillel Yafe Medical Center - Endocrinology dep, Hadera
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center Osteoporosis Center, Jerusalem